CLINICAL TRIAL: NCT00247871
Title: The Prevalence of Panton Valentine Leukocidin, Exfoliative Toxin and Agr Genotypes in Staphylococcus Aureus Nasal Colonization in Vancouver's Eastside Community
Brief Title: Microbiological Characterization and Nasal Carriage Rates of Methicillin Resistant Staphylococcus Aureus (MRSA) in Vancouver Downtown Eastside
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: C05-0193
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Nasal Colonization With MRSA Bacteria
Keywords: MRSA, USA300, CMRSA-10, CMRSA-6, soft tissue abscesses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
We plan to compare data from 300 nasal swab in Vancouver's Downtown Eastside taken in 2001 to data obtained in 2005. The nasal carriage rate of MRSA and the specific characteristic of each MRSA found will be analyzed. A limited amount of associated information will be obtained

DETAILED DESCRIPTION:
MRSA samples will be characterized by pulse field gel electropheresis. An 9 item questionnaire will be administered.

ELIGIBILITY:
Inclusion Criteria:

Patient had a microbiological sample submitted from the emergency department of the study hospital from 2001- 2005 which grew MRSA.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Vancouver's Downtown Eastside
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2005-10-01; Primary Completion 2005-12-01 (Actual); Study Completion 2012-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Reynolds, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada